CLINICAL TRIAL: NCT00924508
Title: A Study to Compare the Efficacy of Triamcinolone 0.1% Cream Occluded With Hydrogel Patch to Triamcinolone 0.1% Cream Without Occlusion in the Treatment of Eczema
Brief Title: Hydrogel Patch for the Treatment of Eczema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of Funding
Sponsor: University of California, San Francisco (Other)
Collaborators: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hydrogel for Eczema
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Eczema
Keywords: eczema; at least 3 patches of eczema
MeSH Terms: conditions — Eczema | interventions — Dental Occlusion; Transdermal Patch; Bandages, Hydrocolloid; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patch + cream, patch alone, cream alone (Experimental): This is a single arm study. Each subject will have 3 target lesions; one treated with TAC 0.1% cream and hydrogel patch (occlusion), the second treated with cream alone, and the third treated with occlusion alone.
  Interventions: Device: hydrogel patch; Drug: Triamcinolone (TAC) 0.1% cream

INTERVENTIONS:
Device: hydrogel patch — occlusion of eczema with a hydrogel patch composed of an adhesive, thin, flexible, hydrogel layer on an impermeable urethane surface.
  Other Names: Occlusion; Patch; Hydrogel
Drug: Triamcinolone (TAC) 0.1% cream — Triamcinolone Acetonide (triamcinolone acetonide cream) is a topical corticosteroid used as anti-inflammatory and antipruritic agent. Each gram of TAC Cream USP, 0.1% contains 1 mg Triamcinolone Acetonide (triamcinolone acetonide cream) in a cream base consisting of cetyl alcohol, glyceryl monostearate, cetyl esters wax, isopropyl palmitate, polysorbate-60, polysorbate-80, propylene glycol and purified water.
  Other Names: Triamcinolone Acetonide cream; TAC cream [United States Pharmacopeia; (USP), 0.1%]

SUMMARY:
The primary objective of this clinical study is to determine whether occlusion of triamcinolone 0.1% cream (TAC) with hydrogel patch improves its efficacy in treating eczema. A secondary objective is to determine whether eczema improves under occlusion with hydrogel patch alone, without TAC.

DETAILED DESCRIPTION:
This will be a 6-week, open label, bilaterally-controlled single center study involving 30 subjects age 13 and older with eczema. The primary objective of this clinical study is to determine whether occlusion of triamcinolone 0.1% cream (TAC) used to treat eczema with hydrogel patch improves its efficacy. A secondary objective is to determine whether eczema improves under occlusion with hydrogel patch alone. All subjects will have 3 target lesions of similar severity followed throughout the study. Patients will apply hydrogel patch alone to the first lesion, TAC 0.1% cream to the second lesion, and TAC 0.1% cream occluded by hydrogel patch to the third lesion. All treatments are twice a day for a maximum of 4 weeks or until lesions are cleared. The modified Eczema Area and Severity Index (EASI) score will be used to evaluate each lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the informed consent form and Health Insurance Portability and Accountability Act (HIPAA) authorization form;
2. Male or female subject at least 12 years of age; subjects under 18 years of age will need parental or official guardian consent.
3. A diagnosis of eczema with at least three lesions no larger than 7 by 7 cm on either the trunk, arms, or legs that would serve as target lesions. The lesions must be wide enough apart so that there is no overlap of hydrogel patches. All three lesions must have at least 5 out of 12 points on the modified EASI scale. Each of the three lesions must have no greater than 1 point difference from each other on the modified EASI score. (If the subject can identify specific eczema lesions that are more pruritic, recalcitrant and/or tend to initiate the itch-scratch cycle, then those lesions will be preferentially selected as the target lesions.)
4. Any additional diagnoses must, in the investigator's opinion, not preclude the subject from safely participating in this study or interfere with the evaluation of the subject's eczema;
5. Subject is able to completely discontinue the use of any medication or therapy (other than study medications) for relief of eczema in the target areas to be treated;
6. Subject is able to completely discontinue the use of any systemic medication or therapy (e.g. oral medications, phototherapy, herbal remedies, or acupuncture) for relief of eczema;
7. Subject must be reliable and mentally competent to complete study measurements;
8. Subject is able to understand and agrees to comply with study requirements, attend study visits, and comply with the restrictions during the study.

Exclusion Criteria:

1. Subjects with exclusively hand, face, foot, and/or groin dermatitis
2. Known hypersensitivity to any component of the test medications;
3. Pigmentation, extensive scarring, or pigmented lesions in affected areas that would interfere with evaluation of efficacy parameters;
4. Clinically infected eczema at baseline.
5. Any evidence of atrophy in the areas selected for treatment with topical corticosteroid;
6. Subjects requiring any other medication (topical or systemic) that may affect the course of the disease during the study period (e.g. oral corticosteroids, immunosuppressants, antibiotics, sedating antihistamines). Inhaled steroids will be permitted.
7. Topical therapies (other than non-prescription emollients) on potential target lesions within one week of starting study treatment;
8. Systemic therapy, phototherapy, or a systemic investigational therapy for eczema within 30 days prior to study entry;
9. Subject is considered unreliable as to medication compliance or adherence to scheduled appointments as determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis Skin and Treatment Center, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible eczema patients from one U.S. clinical site were invited to participate
Pre-assignment Details: Consent was initially obtained from 23 participants, but 3 participants withdrew consent
Groups:
- TAC With Hydrogel Patch, Hydrogel Patch Alone, TAC Alone: This is a single arm study. Each subject had 3 target lesions; one treated with occlusion of lesion by hydrogel patch and 0.1% TAC, the second treated with 0.1% TAC without occlusion, and the third treated with occlusion of eczema lesion by hydrogel patch without TAC.
Period: Overall Study
Arm/Group | TAC With Hydrogel Patch, Hydrogel Patch Alone, TAC Alone
Started | 23
Completed | 20
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | TAC With Hydrogel Patch, Hydrogel Patch Alone, TAC Alone
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (19.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Severity: Percent Change in Mean EASI Score
Description: Percent change in mean EASI score week 0 to week 6: Each lesion was scored using a 12-point modified Eczema Area and Severity Index (EASI) at baseline and 2 weeks after the 4-week treatment period (week6). An experienced evaluator assessed each lesion on the severity of 4 domains, with higher scores indicating more severity: 1) intensity of redness (erythema), 2) thickness (induration, papulation, oedema), 3) scratching (excoriation) and 4) lichenification (lined skin) as as none (0), mild (1), moderate (2) and severe (3). Pictorial and descriptive instructions guided the evaluator in scoring the lesions based on visual appearance.
Time Frame: Baseline, 6 weeks
Population: 3 of 23 enrolled participants withdrew consent and did not provide data for analysis. Each participant had 3 lesions treated in the study, one by each of 3 study treatments.
Measure: Mean (Full Range); unit: percentage change
Units Other Than Participants: Lesions
Groups:
- Hydrogel Patch: Patients were instructed to apply the hydrogel patch over one lesion for 6-8 hours daily. After 4 weeks of occlusion therapy, treatment was discontinued and final evaluation was conducted after a 2-week observation period involving no active therapy.
- TAC 0.1%: Patients were instructed to apply TAC 0.1% twice daily to one lesion. After 4 weeks, treatment was discontinued and final evaluation was conducted after a 2-week observation period involving no active therapy.
- Patch + TAC: Patients were instructed to apply the hydrogel patch over one lesion for 6-8 hours daily and triamcinolone (TAC) 0.1% cream twice daily to one lesion. After 4 weeks of occlusion + TAC treatment, treatment was discontinued and final evaluation was conducted after a 2-week observation period involving no active therapy.
Arm/Group | Hydrogel Patch | TAC 0.1% | Patch + TAC
Number analyzed (Participants) | 20 | 20 | 20
Number analyzed (Lesions) | 20 | 20 | 20
percentage change | -47 [-100 to 17] | -56 [-100 to 0] | -61 [-100 to 17]
Statistical Analysis 1: Comparison: Hydrogel Patch; Baseline and post-treatment comparison; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: TAC 0.1%; Baseline and post-treatment comparison; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Patch + TAC; Baseline and post-treatment comparison; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Number of Adverse Events Associated With Treatment
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: Adverse events
Groups:
- Hydrogel Patch Alone, TAC 0.1%, TAC + Patch: This is a single arm study. Each subject had 3 target lesions; one treated with occlusion of eczema patch with hydrogel and 0.1 % triamcinolone ointment, the second treated with 0.1 % triamcinolone ointment without patch, and the third treated with occlusion of eczema patch without ointment.
  occlusion of eczema patch with hydrogel and 0.1 % triamcinolone ointment, occlusion alone, and ointment alone
Arm/Group | Hydrogel Patch Alone, TAC 0.1%, TAC + Patch
Number analyzed (Participants) | 20
Adverse events | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | TAC With Hydrogel Patch, Hydrogel Patch Alone, TAC Alone
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Due to loss of funding, enrollment was terminated prior to intended accrual of 30 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes